CLINICAL TRIAL: NCT03387072
Title: CIQTP Prolongation : Role and Mechanism in Sudden Cardiac Death
Acronym: IQARE-SCD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0357
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Sudden Cardiac Death
Keywords: Mental stress; Sudden cardiac death; arrhythmias; long QT syndrome
MeSH Terms: conditions — Death, Sudden, Cardiac; Stress, Psychological; Arrhythmias, Cardiac; Long QT Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample (10mL ) for adult patient and teenagers and salivary sample for minor patients (under 12 years of age)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients affected with CIQTP: Patients affected with catecholamine-induced QT prolongation (CIQTP)
  Interventions: Other: Non interventional study
- Healthy relatives of patients affected with CIQTP: Healthy relatives of patients affected with CIQTP identified during the familial screening
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — mental stress test and Blood (or salivary) sample

SUMMARY:
Despite major progress in molecular and phenotypic characterization of primary electrical disorders, many (aborted) sudden cardiac deaths (SCD) occur in young victims without identifiable abnormalities. Investigator recently identified, in 4 families presenting unexplained SCD, a new arrhythmia entity (catecholamine-induced QT prolongation; CIQTP) characterized by normal QT duration at rest but major QT lengthening during mental stress test (MST).

Investigators aim to determine the prevalence of this new phenotype in unexplained SCD and identify its underlying pathophysiological mechanism.

More specifically, investigators aim to:

* determine the prevalence of CIQTP in unexplained SCD and identify new affected families;
* identify the role of mental stress in QT prolongation;
* identify the genetics basis underlying this life threatening disease;
* perform transcriptomic and electrophysiological profiling of induced pluripotent stem cell-derived cardiomyocytes (iPSC-CM) from CIQTP patients to identify putative biomarkers and pathophysiological mechanisms.

MST will be performed, additionally to the conventional screening, in families affected by unexplained SCD or long QT syndrome (LQTS) referred to university hospitals of Nantes, Rennes, Tours and Brest. Relevance of the MST on the different type of LQTS will be evaluated and compared to conventional provocative tests (epinephrine, exercise).

Whole-genome sequencing will first be performed in 3 distantly affected relatives within each of the 4 largest families identified. As previously performed in Nantes, analysis of the shared rare variants will allow identifying gene(s) associated with the disease.

Transcriptomic (high-throughput 3' Digital Gene Expression mRNA sequencing) and electrophysiological (96-well automated optical recordings of action potentials and patch-clamp recordings of ionic currents, using specific ion channel activators and inhibitors) profiling will be performed on iPSC-CMs from 2 affected and one unaffected first-degree relatives of these 4 large families.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is a major cause of death in developed countries. An estimated 40,000 to 50,000 individuals die suddenly each year in France. Most of these deaths involve elderly people and are related to coronary artery disease. However, an estimated 4000 to 5000 individuals between 1 and 45 years of age die suddenly each year in France. SCD often occurs in young victims without identifiable ECG abnormalities and without structural defects. In consequence, most SCD events in the young adult remain unexplained and are classified in an elusive group known as idiopathic ventricular fibrillation (IVF).

Investigator recently identified a new arrhythmic entity (catecholamine-induced QT prolongation; CIQTP) responsible for SCD and characterized by normal QT duration at rest but major QT lengthening during mental stress test. The aim of this translational project is to determine the prevalence of this new phenotype of rare disease in unexplained SCD and identify its underlying pathophysiological mechanism.

The use of mental stress test could be extended to other inherited arrhythmic disease such as long QT syndrome. Given the potential of identification of new affected relatives it may lead to a significant reduction of the risk of sudden cardiac death recurrence in a family.

The main issue of this project is to describe the clinical implication and the pathophysiological mechanism of this new syndrome leading to SCD.

Based on our recent description of this cathecholamine induced QT prolongation, the investigators hypothesize that:

* This syndrome is partly involved in the 60% of undiagnosed familial IVF after complete familial screening7. Indeed, as the baseline ECG is normal without MST, identification of such clinical features may be performed by mental stress test in proband and relatives previously considered as unaffected by inherited arrhythmic disease.
* Mental stress test will help to identify borderline cases of other inherited arrhythmia such as long QT syndrome. Indeed, this inherited arrhythmia is characterised by a genetic-based prolongation of the QT interval observed on the baseline ECG, however more than a third of the patients present with only a slight QT prolongation at baseline. Consequently, they require the use of provocation tests (e.g. exercise test and adrenaline test) to unmask pathological QT prolongation18. The Investigator hypothesize that MST may help to unmask this QT prolongation.
* Based on the autosomal inheritance mode investigator recently described for this disease, investigator hypothesize that this syndrome belongs to the mendelian disorders. Therefore, the investigators propose to apply a familial-based approach to identify the major genes associated with the CIQTP syndrome.

The scope of this project is to describe the clinical implication and the pathophysiological mechanism of this new syndrome leading to sudden cardiac death. More specifically, the investigators aim to:

* determine the prevalence of CIQTP in unexplained SCD and identify new large affected families
* identify the role of mental stress in QT prolongation
* identify associated genes with the disease combining whole genome sequencing and Identity By Descent analysis in large families
* perform transcriptomic and electrophysiological profiling of induced pluripotent stem cell-derived cardiomyocytes (iPSC-CM) from CIQTP patients to identify putative biomarkers and pathophysiological mechanisms.

Based on this translational approach, the investigators aim to describe pathophysiology and clinical implication of CIQTP in sudden cardiac death. The description of this new syndrome using innovative approach such as whole genome sequencing and iPSC-CM profiling may provide a comprehensive and major progress in the field of unexplained SCD. Beyond the identification and the care of newly affected relatives, it may help defining a genetic/pathophysiology based therapy.

The investigators already proved that MST is a highly efficient diagnostic tool to detect this new syndrome, and the investigators believe that it may also help to unmask QT prolongation in silent LQTS mutation carriers. MST has the advantage of being rapid and simple to apply. It could thus be of great interest to uncover familial segregation for unexplained cardiac electrical defects showing autosomal dominant transmission. It could additionally decrease the apparent non-penetrance encountered in LQTS.

Tasks of the project

Task 1: determine the prevalence of CIQTP in unexplained SCD and identify new affected families

Most cases of SCD before the age of 45 remain unexplained and are likely to be due to inherited arrhythmic disease6. After unexplained SCD, all consecutive families referred to Nantes, Rennes, Tours or Brest University Hospitals will be included in the study.

All available clinical proband data will be collected from the referring physicians and relatives. When autopsy is performed, the probands whose diagnosis will be achievable will be excluded from the study.

Familial screening After unexplained SCD before the age of 45, familial screening will be performed in first-degree relatives and then extended to other relatives if positive. When first-degree relatives are not available for screening, it will be performed in more distant relatives.

Clinical screening will include a review of past medical history, clinical examination and baseline ECG. In the absence of diagnosis after this first set of exams, stress test, transthoracic echocardiogram (TTE), sodium channel blocker challenge (SCBC) either with ajmaline (1 mg/kg) or flecainide (2 mg/kg) and an epinephrine test23,24 will be performed. Mental stress test will be additionally performed to unmask QT prolongation with normal baseline ECG 25.

Mental stress test protocol (appendix 2) MST will be performed as follows. Patients will be placed in supine position with no explanation on the course of the test. ECG will be recorded at baseline and permanently during the test. MST will be then performed abruptly according to the patient's level of education (mental arithmetic, geography or names of Disney characters for children) with a requirement for correct and rapid answers. MST will be considered as relevant in the presence of at least a 20 beats-per-minute increase in heart rate. In case of absence of a 20 beats-per-minute increase in heart rate, the test will be considered as non-interpretable unless a significant prolongation of the QTc is identified. MST usually lasts less than 2 minutes. A new ECG will be recorded 30 minutes after the end of the test in an attempt to obtain an ECG trace with the lowest heart rate.

Diagnosis

ECG performed at baseline, during the stress test and during the pharmacological test will be reviewed by two physicians blinded to the clinical and genetic status. All the data will be collected in a core database.

The diagnosis criteria adhered to the guidelines of the latest consensus conference24,26. The investigators will additionally consider a delta QTm > 30 ms during epinephrine or the mental stress test and a delta QTc > 30 ms at 3 min after the stress test, as sufficient for diagnosis of LQTS 27,28.

A minimum interval of 30 minutes between each test will be observed to enable catecholamine clearance. All tests will be performed at least 5 days after interrupting each treatment that could interfere with the tests.

This study is conducted according to European guidelines for clinical and genetic research. Protocol approval will be obtained from institutional ethical committees. Informed written consent will be obtained from each patient who agreed to participate to the clinical and genetic study.

Statistical analysis Statistical analyses will be performed with Social Science® software (IBM Corp., Armonk, New York). Categorical variables will be presented with their numbers and percentages. The chi-square or Fisher exact test (based on expected frequency) will be used to compare categorical variables between groups.

Quantitative variables will be presented as mean ± standard deviation or median (25th; 75th). Analysis of continuous variables will be performed using a t-test or Mann Whitney test based on distribution. Comparisons among families will be performed using intra-familial mean value or median of continuous variable in order to limit the bias toward family size. A two-sided P-value of less than 0.05 will be considered to indicate statistical significance in all tests.

Task 2: identify the role of mental stress in QT prolongation

To identify the role of mental stress in QT prolongation the investigators will additionally enroll positive and negative control groups in Nantes, Rennes, Tours or Brest University Hospitals.

This will consist in the enrolment of consecutive relatives of families affected by long QT syndrome without QT prolongation at baseline. The result of this test will be compared to conventional screening using exercise test and epinephrine test. Thereby, the investigators aim to enroll patient further defined as carriers of the main genetic-based forms of long QT syndrome (LQT1, LQT2 and LQT3, positive control group).

The investigators will additionally enrol a negative control group of healthy patients with normal baseline ECG, no cardiac structural abnormalities and without any medication that could interfere with the MST. This population will consist in relatives of families negative for unexplained SCD screening.

Diagnosis criteria and test protocol will be identical to those defined in task 1.

Three consecutive beats will be used for each measurement and the average value obtained by the two investigators will be taken into account. QT interval will be measured in DII or V5, from the beginning of the QRS complex to the end of the T-wave (defined as the intersection of the tangent of the T-wave and the isoelectric line). U-wave will be excluded from the measurement of the QT interval.

This study is conducted according to European guidelines for clinical and genetic research. Protocol approval will be obtained from institutional ethical committees. Informed written consent will be obtained from each patient who agreed to participate in the clinical and genetic study.

Statistical analyses will be performed with Social Science® software (IBM Corp., Armonk, New York). Comparisons between groups will be performed for each clinical and ECG parameter at baseline and during both tests (mental stress test, exercise test, epinephrine test). Categorical variables will be presented with their numbers and percentages. The chi-square or Fisher exact test (based on expected frequency) will be used to compare categorical variables between groups. Quantitative variables will be presented as mean ± standard deviation or median (25th; 75th). Analysis of continuous variables will be performed using a t-test or Mann Whitney test based on distribution. A two-sided P-value of less than 0.05 will be considered to indicate statistical significance in all tests.

Investigator have already enrolled in Nantes hospital a population of 30 healthy controls and 25 subjects affected with LQTS (LQT1=9 or LQT2=16) but with a resting QTc<480 ms. First results have identified a sensitivity of exercise test, epinephrine test and MST respectively of 60%, 95% and 94% within the families, and 76%, 93% and 92% within the positive controls, for a specificity of 100% reached for every test. This confirms that MST test may be of interest in long QT patients with an absence of clear QT prolongation.

Task 3: identify specific genes associated with the disease

Objective: To identify rare variants in new genes contributing strongly the risk of VF within pedigrees.

Four large IVF families presenting 6 SCD (with 2 resuscitated) and 7 unexplained syncope episodes occurring at young age have been characterized in Nantes. Among them, respectively 9, 10, 11, and 4 family members show a prolonged QT interval after MST and/or another provocative test while all LQTS-associated genes were negative. The description of this new clinical entity has been recently accepted for publication in the Journal of the American College of Cardiology17. The occurrence of VF/SCD or ECG abnormalities in genetically distant individuals within families makes pedigrees highly powerful for genetic studies, since the greater the genetic distance, the less variants the patients will share. Of note additional relatives will be clinically investigated (individual with question mark symbols on pedigrees below) and may increase the power of the genetics study. Previous works of J. Barc and Nantes group demonstrated our capability to lead such ambitious projects and specifically on gene discovery based on familial approach coupled to next generation sequencing.

task3.1: Whole genome genotyping and analysis of the affected family members Aim: Identify a genomic region shared by the affected members.

Genome-wide genotyping on all affected family members will be performed using Axiom Genome-Wide Human Precision Medicine Research Array (PMRA) Plate on Affymetrix GeneTitan® Multi-Channel, instrument available through the genomic core facility of Nantes of our lab. Genomic regions shared by affected family members will be assessed by Identity By Descent (IBD) analysis as previously described. This step is crucial to refine the genome region where the causal variant is located. According the large size of the families the investigators can expect that a relatively small genomic region will come up from this analysis. Attention will be dedicated to potential shared region among families that would indicate a potential common gene.

task3.2: Whole genome sequencing and analysis Aim: identify rare variants among the genomic regions shared by affected family members.

Here the investigators shall carry out genome sequencing in 3 distantly related individuals affected by CIQTP syndrome from each of the 4 pedigrees. Advantages with genome sequencing reside on the absence of capturing and PCR steps, limiting strongly the capture artefacts, the non-covered regions and offering the possibility of uncovering a mutation within an essential regulatory element belonging to the non-coding region. Sequencing will be performed in collaboration with the National Genotyping Center (CEA-CNG). The NGS pipeline follows the recommendations of the Broad Institute GATK "Best Practices" broadinstitute.org/gatk/guide/best-practices.php. Basically, reads are mapped using bwa-mem, Duplicates are removed using picard, GATK is used to realign and recalibrate the reads. The variants are called with HaplotypeCaller and are recalibrated with GATK. The generated VCFs are then annotated with Ensembl Variant Effect predictor. From VCF files and within each pedigree, the investigators shall prioritize variants shared by the 3 affected individuals and contained within shared genomic regions (IBD). From the shared variants the investigators shall focus on rare variants and then filter out variants that are common in the general population (minor allele frequency >0.1%). For this the investigators will use public and in-house exome/genome databases gathering in total about 130 000 exomes and 20 000 genomes such as The gnomAD consortium, 1000Genomes, the Genome of the Netherlands and demographic matched controls specifically from Nantes area (PREGO study-www.vacarme-project.org). This is expected to result in a short-list of few "candidate" variants/genes per family. A bioinformatics prediction of their functional effect will be assessed by the programs SIFT and Polyphen2 to highlight putative malignant variants among those. The investigators will validate all variants identified in such way by Sanger sequencing and investigate their co-segregation with other affected family members in the respective pedigrees. Experience of the genomics and bioinformatics core facility of Nantes of our lab, which are recognized as French national infrastructures in genomics (IBiSA) and bioinformatics (Institut Français de Bioinformatique) coupled to our experience in NGS data managing will assure the feasibility of this Task. Furthermore a large genome sequencing project gathering more than 1000 whole genome (including cardiac patients and individuals from the general population) is on going in our group. Experience from this project will reinforce the efficiency of the task#3 analysis and chance of success.

Task 4: perform transcriptomic and electrophysiological profiling of induced pluripotent stem cell-derived cardiomyocytes from CIQTP patients to identify putative biomarkers and pathophysiological mechanisms

The investigators make the hypothesis that induced pluripotent stem cell-derived cardiomyocytes (iPSC-CMs) generated from CIQPT patients will allow us to identify the global gene expression changes and electrophysiological alterations associated with the disease. For that, the investigators aim at comparing iPSC-CMs generated from members of the 4 families described in task 3. Within each pedigree the investigators will select one "control" healthy subject (not presenting the familial QT prolongation), and 2 CIPQT patients.

Positive LQT control and negative healthy control iPS cell lines have already been generated and studied in Nantes in a context of a previous study on LQT2 demonstrating the feasibility of this task. This will also offer the opportunity to compare CIPQT transcriptomic and electrophysiological signature to LTQ2 ones. For each line, 3 iPS cell clones have been validated: all lines have normal karyotype and meet the current standards for pluripotency. The investigators successfully differentiated the iPS cells into the cardiac lineage, using a recently described method based on temporal modulation of Wnt/ß-catenin signaling using small molecules. Preliminary data suggest that the investigators can generate high purity and efficiency of cardiac differentiation. Regarding the iPS cells from the LQT2 patient, the investigators showed that hERG A561P mutation leads to a trafficking defect that results in reduced IKr current, and consequently e to action potential prolongation and cellular arrhythmias(early afterdepolarizations) .

Upon obtainment and validation of all iPS cell lines, the first step of the project will consist in the identification of the cardiac gene expression profile associated with CIQTP. For that, the investigators will use cardiomyocytes differentiated from control and patient-derived iPS cells (day 28) to perform RNA seq analyses, in collaboration with the Genomics core facility of our lab. The investigators will also perform high-throughput action potential and ionic current analyses using automated patch clamp and optical based (CellOptiq®) techniques under baseline conditions and after drug-induced adrenergic stimulation. All combined, these analyses will provide us with the first identification of the electrophysiological profile associated with CIQTP in human cardiomyocytes. With this analysis, the investigators will be able to link CIQTP-associated altered gene expression program to defective cardiac physiology.

iPSC cardiac differentiation protocols: cells will be cultured on a Matrigel-coated plate and exposed to cardiogenic cytokines: CHIR and IWR-1. Beating colonies appear after about 10 days. After 20 days, cells will be dissociated and reseeded for electrophysiological analyses, 10 days later. Finally, after 28 days of differentiation, beating cells will be collected for RNA seq analysis.

Whole transcriptome sequencing (RNAseq): beating iPSC-CMs at 28 days of 3 differentiation from 2 clones of each iPS cell line will be collected and RNA will be extracted using Macherey-Nagel kit. Presence and quantity of each RNA of the samples will then be assessed using next generation sequencing (Illumina HiSeq technology). Bioinformatics analysis will be performed by the BIRD core facility of our lab.

Ionic current recordings by automated patch clamp: CIQTP's repolarization defects likely reflect dysfunction of specific ionic currents that will be recorded using whole cell patch-clamp: sodium current, INa, calcium current, ICa,L, and potassium currents, IKs and IKr.

Action potential recording: This recording will be performed using 2 techniques.

1. Isolated beating cells will be analyzed using perforated patch-clamp technique with amphotericin B at 37oC. Patch pipettes will be filled with a solution that has an ionic composition similar to the intracellular fluid.
2. Action potential optical recordings will be performed on cardiomyocytes after 28 days of differentiation, with 5 µmol/L di-8-ANEPPS as the voltage-sensitive dye using the CellOptiq® technology (Clyde Biosciences). Cells will be incubated at 37°C, 5% CO2 and 20% O2 during the 2 h-incubation of the dye and during the recording.

ELIGIBILITY:
Inclusion Criteria:

* Relatives seen for a familial screening after an unexplained sudden cardiac death in a young member of their family (<45 years old).
* Patients affected with CIQTP characterized by normal QT duration at rest but major QT lengthening during mental stress test
* Signed consent

Exclusion Criteria:

* Patients who underwent a sudden cardiac death with an identified cause of the decease after an autopsy
* Patients under trusteeship or under guardianship
* Patients who didn't give their consent or who is not able to

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited by the Hereditary or rare heart rhythm disorders reference centre of the Nantes University Hospital, which specialises in the management of patients with sudden death risk pathologies and family screening. The reference centre works in network with the regional competence centres, including the Brest, Rennes and Tours University Hospital Centres.
  Patients will be included in a cardiological consultation or day hospitalization as part of the family screening for sudden death. Family screening is carried out within the usual framework of patient care and in accordance with international recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Number of families diagnosed with a CIQTP syndrome compared to the number of families who underwent a familial screening after a sudden cardiac death | 12 months

SECONDARY OUTCOMES:
Identification of genetics variants involved in the occurrence of CIQTP syndrome | 24 months
gene and ionic current expression modifications between healthy and affected relatives | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste GOURRAUD, Dr, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No